CLINICAL TRIAL: NCT05452512
Title: An Open, Randomized and Parallel-design Exploratory Clinical Trial to Evaluate the Effect of Smart Medication Adherence Monitoring on the Medication Adherence and Blood Vitamin D Concentration
Brief Title: Medication Adherence Monitoring Trial Using Smart Clinical Trial Application and Smart Watch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kim Heejin, Research Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SMART-DRUG-101
Record Dates: First submitted 2022-05-30; First posted 2022-07-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Compliance, Medication
Keywords: smart device; compliance monitoring; vitamin D
MeSH Terms: conditions — Medication Adherence | interventions — Blood Glucose Self-Monitoring; Vitamin D; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self monitoring arm using smart clinical trial application (Sham Comparator): The subjects in this arm will take vitamin D for 3 months and keep track of drug administration using smart clinical trial application (self monitoring).
  Interventions: Other: Self monitoring; Drug: Vitamin D
- Active monitoring using smart watch coupled with self monitoring (Experimental): The subjects in this arm will take vitamin D for 3 months and keep track of drug administration using smart watch and smart clinical trial application (self monitoring).
  Interventions: Other: Self monitoring; Other: Smart watch assisted monitoring; Drug: Vitamin D

INTERVENTIONS:
Other: Self monitoring — Self monitoring using smart clinical trial application
  Other Names: DIARY
Other: Smart watch assisted monitoring — Smart watch-assisted adherence monitoring
  Other Names: SMART WATCH
  Arms: Active monitoring using smart watch coupled with self monitoring
Drug: Vitamin D — Vitamin D self-administration for 3 months
  Other Names: VITAMIN

SUMMARY:
The study will investigate the effect of smart monitoring on medication adherence.

DETAILED DESCRIPTION:
In this study, multiple medication monitoring procedures will be performed: self-reporting, pill counting, smart monitoring and concentration monitoring. Subjects will take vitamin D supplement on the market which enables validated concentration monitoring. The study will last for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-64 years at the consent
* 25(OH) vitamin D < 10 ng/mL
* Not taking vitamin D at the screening
* Fully understood the study procedures

Exclusion Criteria:

* Hypercalciuria, sarcoidosis
* Clinically significant hypersensitivity reaction to Vitamin D
* History of or current kidney stone
* One of the following findings:

  1. Serum calcium level > upper limit of normal
  2. Estimated glomerular filtration rate < 60 mL/min/1.73m^2
* Galactose intolerance, Lapp lactase deficiency, Glucose-galactose malabsorption
* Unable to use smart clinical trial application or smart watch
* Expected to take vitamin D from 4 weeks before the first administration and until the last administration

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
The percentage of prescribed doses taken | 3 months
  Percentage of doses taken
The percentage of days with correct dosing | 3 months
  Taking adherence

SECONDARY OUTCOMES:
The percentage of days with correct dosing window | 3 months
  Timing adherence
Days without medication intake during a time period longer than 24 h | 3 months
  Drug holiday
Mean difference between administration time point and the mode of administration time point | 3 months
  Timing distribution index
Sum of deviations divided by the number of days | 3 months
  Concurrence of medication adherence records
Serum concentration of vitamin D | 3 months (Day 1, 15, 29, 43, 57, 71, 85)
  Vitamin D concentration

CONTACTS AND LOCATIONS:
Overall Officials: Heejin Kim, PhD, Principal Investigator — Seoul National University Hospital Clinical Trial Center
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No